CLINICAL TRIAL: NCT00696371
Title: PET Imaging of Peripheral Benzodiazepine Receptors Using [11C](R)-PK 11195 and [11C]PBR28
Brief Title: PET Imaging of Peripheral Benzodiazepine Receptors
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080158; 08-M-0158
Record Dates: First submitted 2008-06-11; First posted 2008-06-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-08-19

CONDITIONS: Healthy
Keywords: Neuroinflammation; PBR28; PET Imaging; Health Volunteer; HV
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will use positron emission tomography (PET) to measure a receptor in the brain that is involved in inflammation. It will test two radioactive chemicals used in the procedure to see if the newer chemical, [(11)C]B, is as good or better than the older one, [(11)C]A, for measuring brain inflammation.

Healthy volunteers 18 years of age and older may be eligible for this study. Participants undergo an evaluation, [(11)C]A PET scan, [(11)C]B PET scan and magnetic resonance imaging (MRI), as follows:

Evaluation

Medical history and physical examination, blood and urine tests

PET scans

* [(11)C]A scan. A catheter (plastic tube) is placed in an arm vein for injection of the [(11)C]A isotope. Some patients also have a catheter placed in an artery in the wrist to collect arterial blood samples during the scan. Subjects then lie on the scanner bed and a special mask is fitted to the head to help keep the subject s head still during the procedure. Following an 8-minute scan to calibrate the scanner, the [(11)C]A is injected into the catheter in the vein and pictures are taken that show where chemicals related to inflammation are present. The procedure takes about 2.5 hours.
* [(11)C]B scan. The procedure is the same as above for [(11)C]A, except the isotope used is [(11)C]B.

MRI scan.

This test uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The subject lies on a table that can slide in and out of the scanner (a metal cylinder), wearing earplugs to muffle loud noises that occur during the scan.

...

DETAILED DESCRIPTION:
Objective:

In response to brain inflammation, microglia over-express the peripheral benzodiazepine receptor (PBR). Although peripheral organs such as the heart and kidney express PBR constitutively, the brain normally expresses PBR in low numbers. Increased PBR density in the brain therefore signifies a change from a normal state to an active, inflammatory state. Positron emission tomography (PET) imaging can quantify PBR density in vivo using radioligands that bind to PBR sites. One PBR-selective radioligand, [(11)C](R)-PK 11195, has been used to identify areas of brain inflammation in patients with various neurological diseases. Unfortunately, [(11)C](R)-PK 11195 has several limitations, including low specific signal. A recently developed radioligand, [(11)C]PBR28, has higher specificity than [(11)C](R)-PK 11195 for PBR in animal studies. No study to date has compared [(11)C]PBR28 to [(11)C](R)-PK 11195 in human subjects.

In early clinical studies using [(11)C]PBR28, 4 of 32 healthy human subjects had complete absence of radioligand binding, even in peripheral organs that constitutively express PBR. One of these non-binders had specific binding of PBR28 on an in vitro assay using peripheral lymphocytes. We do not know why some subjects have [(11)C]PBR28 binding while others do not. We also do not know why one non-binder had positive in vitro binding and negative in vivo binding on PET imaging. No study has reported absent binding with [(11)C](R)-PK 11195. In order to better understand the phenomenon of non-binding, we need to obtain [(11)C](R)-PK 11195 PET scans in subjects that are [(11)C]PBR28 non-binders.

Study Population:

This protocol will study a total of 30 healthy human volunteers.

Design:

Fifteen subjects will undergo PET imaging with [(11)C]PBR28 and [(11)C](R)-PK 11195 using arterial blood sampling for fully quantitative image analysis. These subjects may have dedicated brain PET imaging or whole body PET imaging.

Fifteen subjects will undergo PET imaging with [(11)C]PBR28 and [(11)C](R)-PK 11195 without arterial blood sampling. These subjects will have whole body PET imaging.

All subjects will have in vitro PBR28 binding assays performed.

<TAB>

Outcome Measures:

Our primary outcome measures will be the distribution volume and time stability of each radioligand. We also wish to determine if subjects with absent [(11)C]PBR28 binding also have absent [(11)C](R)-PK 11195 binding. The presence or absence of [(11)C]PBR28 and [(11)C](R)-PK 11195 binding will be evaluated in brain and in peripheral organs. Lastly, we will measure in vitro binding of PBR28 by performing binding assays using peripheral blood cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must be healthy and at least 18 years of age.

EXCLUSION CRITERIA:

* Current psychiatric disease, substance abuse or severe systemic disease based on history and physical exam.
* Laboratory tests with clinically significant abnormalities.
* Prior participation in other research protocols or clinical care in the last year such that radiation exposure, including that from this protocol, would exceed the guidelines set by the Radiation Safety Committee (RSC).
* Pregnancy or breast feeding.
* Positive result on urine screen for illicit drugs.
* Subjects who cannot lie on their back for extended periods of time.
* Subjects with significant claustrophobia who cannot tolerate an MRI scan.
* Subjects with cardiac pacemakers or metal in their bodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06-06; Study Completion 2014-08-19

PRIMARY OUTCOMES:
The first goal of this study is to compare [11C]PBR28 and [11C](R)-PK 11195 as radioligands in the measurement of PBR in healthy human subjects. Our primary outcome measures will be the distribution volume and time stability of each radioligand.

SECONDARY OUTCOMES:
The second goal is to identify non-binders, that is, subjects that do not demonstrate any binding to [11C]PBR28.

CONTACTS AND LOCATIONS:
Overall Officials: William C Kreisl, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anholt RR, De Souza EB, Oster-Granite ML, Snyder SH. Peripheral-type benzodiazepine receptors: autoradiographic localization in whole-body sections of neonatal rats. J Pharmacol Exp Ther. 1985 May;233(2):517-26. PMID 2987488
- [Background] Banati RB, Myers R, Kreutzberg GW. PK ('peripheral benzodiazepine')--binding sites in the CNS indicate early and discrete brain lesions: microautoradiographic detection of [3H]PK11195 binding to activated microglia. J Neurocytol. 1997 Feb;26(2):77-82. doi: 10.1023/a:1018567510105. PMID 9181482
- [Background] Banati RB, Newcombe J, Gunn RN, Cagnin A, Turkheimer F, Heppner F, Price G, Wegner F, Giovannoni G, Miller DH, Perkin GD, Smith T, Hewson AK, Bydder G, Kreutzberg GW, Jones T, Cuzner ML, Myers R. The peripheral benzodiazepine binding site in the brain in multiple sclerosis: quantitative in vivo imaging of microglia as a measure of disease activity. Brain. 2000 Nov;123 ( Pt 11):2321-37. doi: 10.1093/brain/123.11.2321. PMID 11050032